CLINICAL TRIAL: NCT00584311
Title: MRI and Ultrasound Findings in Patients With Gout and Normal Plain Radiographs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Responsible Party: John D. Carter, M.D., University of South Florida
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 6123-G62368; 6123-G62368
Record Dates: First submitted 2007-12-20; First posted 2008-01-02 (Estimated); Last update posted 2008-06-09 (Estimated); Status verified 2008-06

CONDITIONS: Gout
MeSH Terms: conditions — Gout | interventions — Magnetic Resonance Spectroscopy; High-Energy Shock Waves

ARMS (1):
- 1 (Experimental): All patients (with no structural damage on the plain x-ray) will receive a MRI and Ultrasound (US) of their most involved joint and an asymptomatic joint.
  Interventions: Other: MRI and Ultrasound

INTERVENTIONS:
Other: MRI and Ultrasound — MRI and US of the joint

SUMMARY:
Radiographic imaging plays a key role in managing the long-term effects of hyperuricemia on the skeletal system. Two of the accepted indications for prophylactic urate-lowering drugs in patients with hyperuricemia are gouty tophi and erosions. While much data exist on the plain radiographic changes that are seen in patients with chronic gout, far less is known about the changes seen on other imaging modalities, such as magnetic resonance imaging (MRI) and ultrasound (US). Further, there is very little data on the MRI and US appearance of asymptomatic joints in patients with hyperuricemia and symptomatic gout.

There is vast emerging data to suggest that MRI and US are much more sensitive than plain radiographs at detecting the early stigmata of rheumatoid arthritis (RA). Indeed, these imaging devices have revolutionized the treatment of RA, for the earlier detection of the skeletal changes of RA often mandates more aggressive therapy. These same changes would often be missed by plain radiographs.

It is our hypothesis that MR imaging and US will detect the skeletal changes that are typical of gout much sooner than would plain radiography. We also hypothesize that these same imaging techniques will be able to detect signs of hyperuricemic silent deposition in asymptomatic joints of patients with symptomatic gout in other joints. As was the case with RA, the expected results of this study would mandate more aggressive therapy of both gout and hyperuricemia.

Our primary aim of this proposal would be accomplished by studying patients with known gout and normal plain radiographs. Each patient would have their most frequently involved joint (index joint) analyzed by MRI and US to evaluate for any destructive changes (erosions or tophi with cortical damage). Any signs that may portend future joint destruction such as synovial pannus, bone marrow edema, soft tissue edema, or joint effusions will also be documented. In order to demonstrate the effects of hyperuricemic silent deposition, an asymptomatic joint from these same patients will be studied using these same imaging techniques. Any evidence of erosions, tophi, synovial pannus, bone marrow or soft tissue edema, or joint effusions will be recorded. By demonstrating destructive, or potentially destructive, skeletal changes in the index joint or asymptomatic joint of a significant number of patients, we will show that patients who are left untreated on the basis of normal plain radiographs are likely to already have skeletal damage.

ELIGIBILITY:
Inclusion Criteria:

* Known history of gout

Exclusion Criteria:

* History of any other inflammatory arthritis (ex. rheumatoid arthritis, psoriatic arthritis)
* History of another crystal induced arthritis (ex. pseudogout)
* Any contraindication to receiving an MRI (ex. pacemaker)
* Allergy to gadolinium contrast dye
* Inability to give informed consent
* Pregnant women
* Erosive changes on initial screening x-ray of index joint
* Serum Creatinine > 1.8 mg/dL at screening visit

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2007-06; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is presence or absence of skeletal damage (on either MRI or US). The data will then be analyzed in the same fashion but by MRI and US independently. | 2 weeks

SECONDARY OUTCOMES:
The presence of erosions, tophi with cortical erosions, tophi without cortical erosions, bone marrow edema/reactive changes, soft tissue edema/swelling, synovial pannus, and joint effusions | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: John D. Carter, M.D., Principal Investigator — University of South Florida
Locations (1):
- University of South Florida, Tampa, Florida, United States